CLINICAL TRIAL: NCT00655616
Title: A Proof-of-concept Study to Evaluate the Benefit From add-on Therapy With Montelukast Versus Salmeterol in Children With Asthma Carrying the Arg/Arg-16 beta2-receptor Genotype
Brief Title: Add-on Salmeterol Versus Montelukast in Arg/Arg-16 Asthmatics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Ms Fiona Hogarth, University of Dundee
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sm2006msd01
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2009-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Salmeterol Xinafoate; montelukast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): The active comparator arm consists of Flixotide® (fluticasone propionate) via accuhaler (Diskus) dry powder inhaler device as per current inhaled steroid dose plus oral montelukast
  Interventions: Drug: Salmeterol, Montelukast
- 2 (Placebo Comparator): The placebo comparator arm consists of Seretide® (salmeterol plus equivalent dose of fluticasone) via accuhaler dry powder inhaler device as per current inhaled steroid dose plus placebo for montelukast
  Interventions: Drug: Montelukast Placebo

INTERVENTIONS:
Drug: Montelukast Placebo — Seretide 100 Accuhaler 1 dose twice daily plus 1 tablet daily of placebo montelukast
  Seretide 250 Accuhaler 1 dose twice daily plus 1 tablet daily of placebo montelukast
  Seretide 500 Accuhaler 1 dose twice daily plus 1 tablet daily of placebo montelukast
  Doses of montelukast or placebo: up to 6 years 4 mg once daily; 6-14 years 5 mg once daily; 15 years and above 10 mg once daily
  Arms: 2
Drug: Salmeterol, Montelukast — Flixotide Accuhaler 50 micrograms per blister, 1 blister dose twice daily plus 1 tablet daily of montelukast
  Flixotide Accuhaler 100 micrograms per blister; 1 blister dose twice daily plus 1 tablet daily of montelukast
  Flixotide Accuhaler 250 micrograms per blister; 1 blister dose twice daily plus 1 tablet daily of montelukast
  Flixotide Accuhaler 500 micrograms per blister; 1 blister dose twice daily plus 1 tablet daily of montelukast
  Doses of montelukast or placebo: up to 6 years 4 mg once daily; 6-14 years 5 mg once daily; 15 years and above 10 mg once daily
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether patients with asthma who carry a genotype associated with adverse outcomes with long-acting beta-2 agonists like salmeterol show greater benefit from the use of an asthma drug that works via alternative pathways like montelukast.

DETAILED DESCRIPTION:
Background/Rationale:

The presence of the homozygous Arg/Arg genotype at position 16 of the β2-receptor (prevalence 15-17% in UK/US populations) confers relative protection against down-regulation by endogenous catecholamines, making individuals susceptible to down-regulation and desensitization by regular exogenous β2-agonists and thereby negating the benefits from the regular use of short and long acting β2-agonists in adults with asthma. We found that, in the children receiving salmeterol, the adjusted odds ratio showed a 9 fold (p=0.003) greater risk of school absences due to asthma in the Arg/Arg group in comparison to the Gly16 carriers, with an unadjusted odds ratio of 6 (p=0.009). In the cohort not receiving salmeterol, there was no evidence of any genotype-dependent increases in school absences due to asthma (odds ratio=1). In addition, the Arg/Arg children on salmeterol had a significantly increased risk of extended school absence of over 1 week from asthma with an adjusted odds ratio of 6 (p= 0.019).

Currently, British Thoracic Society/Scottish Intercollegiate Guidelines Network recommendations suggest the use of regular long-acting β2-agonists as add on therapy in children with asthma who are inadequately controlled on inhaled steroids. The guidelines suggest the use of leukotriene antagonists (e.g. montelukast) if a combination of inhaled salmeterol and inhaled steroids fail to control symptoms.

There are 1 million children with asthma in the UK. 150,000-170,000 children carry the Arg/Arg-16 genotype.

The Arg/Arg-16 children with asthma may constitute a significant population that is likely to show better asthma control with a leukotriene antagonist in comparison to long-acting β2-agonists. We have already demonstrated that school absences constitute a suitable primary outcome measure for the testing of this hypothesis.

Hypothesis:

Children with asthma carrying the Arg/Arg-16 genotype on step 2 of the BTS guidelines (inhaled steroids plus salbutamol according to need) have fewer school absences over a period of 1 year on oral montelukast compared to inhaled salmeterol

Objectives:

To perform a randomized controlled trial (parallel design) of oral montelukast versus inhaled salmeterol on children with a history of school absences/hospital admissions due to asthma over the past year using school absences from asthma over a period of 1 year as the primary outcome

Treatment Groups and Duration:

Inclusion/exclusion criteria- All children and adolescents (5-18 years) with asthma in Tayside (Scotland) known (a) to carry the Arg/Arg-16 genotype and (b) currently on inhaled steroids and (c) inhaled bronchodilators according to need will be telephoned or contacted through home visits to establish if they have had (a) any school absences from asthma or (b) out-of-hours visits to GP/hospital visits or admissions due to asthma over the previous 12 months. The presence of serious respiratory or multi-system disease (e.g. cystic fibrosis, cancer under current treatment) will constitute exclusion criteria for the study. All patients fulfilling the above inclusion and exclusion criteria will be invited to participate in the study.

Plan for each visit - First visit: (a) Documentation of patient details (b) Baseline spirometry; (c) Exhaled nitric oxide measurements (d) Respiratory quality-of-life (Juniper); (e) Saliva sample for eosinophilic cationic protein (f) discontinuation of current asthma medication for the period of the study; (g) randomization to receive either (a) Flixotide (fluticasone) as per current inhaled steroid dose (therapeutic ratio of 2:1 for beclomethasone / budesonide versus fluticasone) plus oral montelukast; or (b) Seretide (salmeterol plus equivalent dose of fluticasone) plus placebo for montelukast for a period of 1 year.

2nd -5th visits, month 3, 6, 9: 3-monthly spirometry, exhaled nitric oxide, saliva for eosinophilic cationic protein, document school absences for asthma, hospital admissions/hospital or out-of-hours GP visits over the 3-month period.

Month 12: end of study - spirometry, exhaled nitric oxide, saliva for eosinophilic cationic protein, document school absences for asthma, hospital admissions/hospital or out-of-hours GP visits over final 3-month period, measure quality-of-life.

Physical monitoring of compliance will be performed by using inhalers provided with counters and tablet dispensers that allow counting of number used.

Doses and dosage regimens:

The following doses and dosage regimens will be used for the study Seretide 100 Accuhaler 1 dose twice daily plus 1 tablet daily of placebo montelukast Seretide 250 Accuhaler 1 dose twice daily plus 1 tablet daily of placebo montelukast Seretide 500 Accuhaler 1 dose twice daily plus 1 tablet daily of placebo montelukast Flixotide Accuhaler 50 micrograms per blister, 1 blister dose twice daily plus 1 tablet daily of montelukast Flixotide Accuhaler 100 micrograms per blister; 1 blister dose twice daily plus 1 tablet daily of montelukast Flixotide Accuhaler 250 micrograms per blister; 1 blister dose twice daily plus 1 tablet daily of montelukast Flixotide Accuhaler 500 micrograms per blister; 1 blister dose twice daily plus 1 tablet daily of montelukast Doses of montelukast or placebo: upto 6 years 4 mg once daily; 6-14 years 5 mg once daily; 15 years and above 10 mg once daily.

Rescue medication: Subjects will be advised treatment with inhaled salbutamol 200 to 1000 micrograms via metered dose inhaler and volumatic device, if cough, breathlessness, increasing symptoms on exercise, or other symptoms of asthma occur. The dose will be advised to be repeated once every four to six hours. The regimen will be advised to be continued for 3-4 days, and up to a week, in case of persistence of symptoms. The research nurse conducting the study will ensure that the subject has an adequate supply of salbutamol via metered dose inhaler and large volume spacer (volumatic) at the start of the study. This will be confirmed at each visit.

Key Efficacy Parameters:

1. Primary outcome: Oral montelukast is associated with reduced school absences in comparison to inhaled salmeterol over a period of 1 year in Arg/Arg-16 asthmatic children
2. Secondary outcomes that will also be tested:

   * Oral montelukast is associated with reduced out-of hours visits/hospital visits or admissions in comparison to inhaled salmeterol over a period of 1 year
   * Oral montelukast is associated with a reduction in airway resistance in comparison to inhaled salmeterol over a period of 1 year
   * Oral montelukast is associated with reduced exhaled nitric oxide levels in comparison to inhaled salmeterol over a period of 1 year
   * Oral montelukast is associated with reduced salivary eosinophilic cationic protein levels in comparison to inhaled salmeterol over a period of 1 year
   * Oral montelukast is associated with improved asthma specific quality-of-life in comparison to inhaled salmeterol over a period of 1 year
   * Oral montelukast is associated with improved morning peak expiratory flow rate in comparison to inhaled salmeterol over a period of 1 year

ELIGIBILITY:
Inclusion Criteria:

All children and adolescents (5-18 years) with asthma in Tayside (Scotland) known:

* To carry the Arg/Arg-16 genotype and
* Currently on inhaled steroids and
* Inhaled bronchodilators according to need will be telephoned or contacted through home visits to establish if they have had:

  * Any school absences from asthma or
  * Out-of-hours visits to GP/hospital visits or admissions due to asthma over the previous 12 months.

Exclusion Criteria:

* The presence of serious respiratory or multi-system disease (e.g. cystic fibrosis, cancer under current treatment)

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2007-08; Primary Completion 2009-08 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Oral montelukast is associated with reduced school absences in comparison to inhaled salmeterol over a period of 1 year in Arg/Arg-16 asthmatic children | Every 3 months

SECONDARY OUTCOMES:
Oral montelukast is associated with improved asthma specific quality-of-life in comparison to inhaled salmeterol over a period of 1 year | Every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Somnath Mukhopadhyay, FRCPCH,PhD, Principal Investigator — University of Dundee
Locations (1):
- Maternal and Child Health Sciences, Ninewells Hospital and Medical School, Dundee, Tayside, United Kingdom

REFERENCES:
- [Background] Palmer CN, Lipworth BJ, Lee S, Ismail T, Macgregor DF, Mukhopadhyay S. Arginine-16 beta2 adrenoceptor genotype predisposes to exacerbations in young asthmatics taking regular salmeterol. Thorax. 2006 Nov;61(11):940-4. doi: 10.1136/thx.2006.059386. Epub 2006 Jun 13. PMID 16772309
- [Derived] Lipworth BJ, Basu K, Donald HP, Tavendale R, Macgregor DF, Ogston SA, Palmer CN, Mukhopadhyay S. Tailored second-line therapy in asthmatic children with the Arg(16) genotype. Clin Sci (Lond). 2013 Apr;124(8):521-8. doi: 10.1042/CS20120528. PMID 23126384